CLINICAL TRIAL: NCT07041125
Title: Ablation With FARAPULSE and Left Atrial Appendage Closure With Watchman for Integrated Management of Atrial Fibrillation)
Brief Title: Concomitant LAAC/AF Ablation (Watchman FLX Pro)
Status: Recruiting | Type: Observational
Sponsor: Heart Rhythm Clinical and Research Solutions, LLC (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ALIGN-AF
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: PFA Ablation and LAAC Procedures
Keywords: AF ablation; FARADRIVE™; Watchman FLX Pro

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Combining LAAC and PFA ablation procedures: AF ablation and LAAC procedures are performed per operators' standard practice. AF ablation will include PVI. Additional right or left atrial ablations are per investigators' discretions. Both AF ablation and LAAC procedures may be performed with ICE or TEE. Assessment of LAAC peri-device leaks and device-related thrombi at 45-90 days may be performed with TEE or cardiac computed tomography angiography (CCTA).
  Interventions: Device: Watchman FLX™ Pro device.

INTERVENTIONS:
Device: Watchman FLX™ Pro device. — Patients eligible for the main DISRUPT-AF Registry with a planned concomitant LAAC procedure using the Watchman FLX™ Pro device.

SUMMARY:
This sub-study is a prospective/retrospective, non-randomized, observational, comparative cohorts study, embedded in and expanding on the infrastructure of a real-world AF ablation registry DISRUPT-AF (NCT06335082).

DETAILED DESCRIPTION:
The prospective arm of the sub-study is intended to enroll 120 subjects indicated for PFA and Watchman in up to 20 US sites within the framework of the DISRUPT-AF registry. Subjects will be screened for eligibility to participate in concomitant PFA ablation for AF and LAAC by Watchman FLX Pro device in a single procedure. Both PVI and LAAC procedures are performed per SOC. In general, percutaneous catheterization will be initially established using FARADRIVE™ steerable sheath for ablation treatment of AF using the FARAWAVE Catheter per instruction for use (IFU) of the device and operator's standard practice. AF ablation will include PVI. Additional right or left atrial ablations are per investigators' discretions. After AF ablation, the FARAWAVE Catheter will be withdrawn. The FARADRIVE™ steerable sheath will be replaced with Watchman FLX deployment sheath. Deployment of Watchman FLX Pro device to LAA to achieve LAAC will follow the standard practice of the care and IFU of the device. Patients will be followed up at 45-90 days for LAAC implant assessment and at 3, 6, and 12 months for arrhythmia recurrence assessment

ELIGIBILITY:
Inclusion Criteria: All inclusion criteria of the main DISRUPT-AF registry will apply. In addition, patients included in this sub study must meet the additional inclusion criteria below:

* Patients who are determined by physicians to be eligible for LAAC
* Patients whose LAAC with Watchman FLX Pro procedures are performed concomitant following AF ablation procedure
* Willing and able to provide additional informed consent to the sub-study (unless waiver of consent is obtained)

Exclusion Criteria: All exclusion criteria of the main DISRUPT-AF registry will apply. In addition, patients included in this sub study have the additional exclusion criteria below:

-Patients who are participating in other DISRUPT-AF sub-studies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients eligible for the main DISRUPT-AF Registry with a planned concomitant LAAC procedure using the Watchman FLX™ Pro device
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
The occurrence of events between the time of implant and within 7 days following the procedure | 12 months
  AF ablation safety will be compared between the concomitant procedures and standalone AF ablation cohort. and LAAC procedure safety will be compared between the concomitant procedures and standalone LAAC cohort.

SECONDARY OUTCOMES:
LAAC success and late-onset safety | 12 months
  45-90 days leaks around LAAC device, 45-90 days device-related thrombus and

OTHER OUTCOMES:
Procedural efficiency: | 12 months
  Number of transseptal crossings, Total procedure time of concomitant, Relative difference in procedure time of stand-alone PFA procedure timevs. concomitant PFA

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Arrhythmia Institute at Grandview, Birmingham, Alabama
  - Arrhythmia Center of South Florida, Delray Beach, Florida
  - Ascension St. Vincent's Jacksonville, Jacksonville, Florida
  - HCA Research Institute- Mercy Hospital, Miami, Florida
  - Ascension St Vincent -Indianapolis Ascension Health, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Heart & Vascular Institute, Louisville, Kentucky
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - St, Mark's Hospital, Salt Lake City, Utah
  - Chippenham Hospital), Richmond, Virginia